CLINICAL TRIAL: NCT00977431
Title: Phase I, Open Label Trial to Explore Safety of Combining BIBW 2992 and Radiotherapy With or Without Temozolomide in Newly Diagnosed GBM
Brief Title: Open Label Trial to Explore Safety of Combining Afatinib (BIBW 2992) and Radiotherapy With or Without Temozolomide in Newly Diagnosed Glioblastoma Multiform
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200.38; 2008-007284-17 (EudraCT Number)
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Radiotherapy; Afatinib

ARMS (2):
- Regimen U (Experimental): BIBW2992 + Radiotherapy
  Interventions: Procedure: Radiotherapy; Drug: BIBW2992
- Regimen M (Experimental): BIBW2992 + Temozolomide + Radiotherapy
  Interventions: Drug: Temozolomide; Drug: BIBW2992; Procedure: Radiotherapy

INTERVENTIONS:
Drug: Temozolomide — During RT: 75 mg/m2 daily , 4 weeks after RT: given days 1 to 5 of 28 day cycles (150 mg/m2 in cycle 1, 200 mg/m2 in cycle 2 up to cycle 6)
  Arms: Regimen M
Procedure: Radiotherapy — Day 1 to day 42
  Arms: Regimen U
Drug: BIBW2992 — Escalating dose cohorts during Radiotherapy(RT) period, fixed dose after RT
  Arms: Regimen M
Procedure: Radiotherapy — Day 1 to day 42
  Arms: Regimen M
Drug: BIBW2992 — Escalating dose cohorts during Radiotherapy(RT) period , fixed dose after RT
  Arms: Regimen U

SUMMARY:
This study is a phase I, open label trial to determine the Maximum Tolerated Dose (MTD), safety, pharmacokinetics, and efficacy of BIBW 2992 (an epidermal growth factor receptor(EGFR)inhibitor) to be used in combination with:

* radiotherapy alone (in patients with an unmethylated (functioning) MGMT gene regulator) or
* radiotherapy and Temozolomide (in patients with a methylated (silenced) O6-methylguanine-DNA methyltransferase gene (MGMT) to treat newly diagnosed patients with Grade IV Glioblastoma (primary brain cancer).

ELIGIBILITY:
Inclusion criteria:

1. Histologically-confirmed WHO Grade IV newly diagnosed malignant glioma.
2. Proven MGMT gene promoter methylation status
3. Available early postoperative Gd-enhanced MRI (within 72 hours after initial surgery). In case a patient did not perform a Gd-enhanced MRI within 72 hours post surgery, a Gd-MRI is to be performed prior to start of study treatment.
4. Age more or equal to 18 years and less than 70 years at entry
5. Karnofsky Performance Scale (KPS) more or equal to 70%
6. Patients receiving corticosteroids have to receive a stable or decreasing dose for at least 14 days before start of treatment.
7. Written informed consent that is consistent with local law and ICH- Good Clinical Practice (GCP) guidelines.

Exclusion criteria:

1. Less than two weeks from surgical resection or other major surgical procedure at start of treatment.
2. Planned surgery for other diseases
3. Placement of Gliadel® wafer at surgery.
4. Prior or planned radiotherapy of the cranium including brachytherapy and/or radiosurgery for GBM.
5. Treatment with other investigational drugs; participation in another clinical study including exposure to the investigational product within the past 4 weeks before start of therapy or concomitantly with this study.
6. Active infectious disease requiring intravenous therapy.
7. Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
8. Gastrointestinal disorders that may interfere with the absorption of the study drug or chronic diarrhoea.
9. Patients with known pre-existing interstitial lung disease
10. Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the protocol.
11. Patient is less than 3 years free of another primary malignancy except: if the other primary malignancy is either not currently clinically significant or does not require active intervention (such as a basal cell skin cancer or a cervical carcinoma in situ). Existence of any other malignant disease is not allowed.
12. Cardiac left ventricular function with resting ejection fraction less than 50%.
13. Absolute neutrophil count (ANC) less than 1500/mm3.
14. Platelet count less than 100,000/mm3.
15. Bilirubin greater than 1.5 x upper limit of institutional norm.
16. Aspartate amino transferase (AST) greater than 3 x upper limit of institutional norm.
17. Serum creatinine greater than 1.5 x upper limit of institutional norm.
18. Patients who are sexually active and unwilling to use a medically acceptable method of contraception.
19. Pregnancy or breast-feeding.
20. Patients unable to comply with the protocol.
21. Known or suspected active drug or alcohol abuse.
22. Known hypersensitivity to BIBW 2992 or the excipients of any of the trial drugs.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-09-17 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (5):
- United Kingdom (5):
  - Addenbrooke's Hospital, Cambridge
  - Ninewells Hospital & Medical School, Dundee
  - Beatson West of Scotland Cancer Centre, Glasgow
  - The Christie Hospital, Manchester
  - The Royal Marsden Hospital, Sutton

REFERENCES:
- [Derived] Saran F, Welsh L, James A, McBain C, Gattamaneni R, Jefferies S, Harris F, Pemberton K, Schaible J, Bender S, Cseh A, Brada M. Afatinib and radiotherapy, with or without temozolomide, in patients with newly diagnosed glioblastoma: results of a phase I trial. J Neurooncol. 2021 Dec;155(3):307-317. doi: 10.1007/s11060-021-03877-6. Epub 2021 Nov 17. PMID 34787778

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is phase I, open-label, non-randomised, uncontrolled dose-escalation trial using a rule-based 3+3 design and patient stratification to explore safety of combining afatinib and radiotherapy with or without temozolomide in newly diagnosed Glioblastoma multiforme (GBM)
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended a specialist sites which ensured that they met all strictly implemented inclusion/exclusion criteria. Patients were not to be entered to trial if any one of the specific entry criteria was violated.
Groups:
- Afatinib 20 Milligram, Radiotherapy + Temozolomide - Regimen M: Patients were administered Afatinib 20 milligram (mg) film-coated tablet once daily orally plus radiotherapy (RT) i.e. focal radiation at a dose of 2 Gray per fraction on 5 days per week for 6 weeks (RT phase) (total dose of 60 Gray (Gy)) plus Temozolomide (TMZ) 75 milligrams per square meter (mg/m2) capsules continuous daily oral dosing. In the maintenance phase after RT, patients stopped TMZ for 4 weeks and restarted TMZ at 150 mg/m2 in cycle 1 and 200 mg/m2 in cycles 2 to 6 on days 1 to 5 of 28-day treatment cycles. Patients were administered Afatinib 40 milligram (mg) film-coated tablet once daily after RT. Dose reductions of Afatinib were allowed if 40 mg or 30 mg were not tolerated. The treatment duration was until tumour progression or occurrence of undue adverse reactions, whichever occurred first.
- Afatinib 30 mg, Radiotherapy + Temozolomide - Regimen M: Patients were administered Afatinib 30 mg film-coated tablet once daily orally plus radiotherapy (RT) i.e. focal radiation at a dose of 2 Gray per fraction on 5 days per week for 6 weeks (RT phase) (total dose of 60 Gray) plus Temozolomide 75 milligrams per square meter (mg/m2) capsules continuous daily oral dosing. In the maintenance phase after RT, patients stopped TMZ for 4 weeks and restarted TMZ at 150 mg/m2 in cycle 1 and 200 mg/m2 in cycles 2 to 6 on days 1 to 5 of 28-day treatment cycles. Patients were administered Afatinib 40 milligram (mg) film-coated tablet once daily after RT. Dose reductions of Afatinib were allowed if 40 mg or 30 mg were not tolerated. The treatment duration was until tumour progression or occurrence of undue adverse reactions, whichever occurred first.
- Afatinib 40 mg, Radiotherapy + Temozolomide - Regimen M: Patients were administered Afatinib 40 mg film-coated tablet once daily orally plus radiotherapy (RT) i.e. focal radiation at a dose of 2 Gray per fraction on 5 days per week for 6 weeks (RT phase) (total dose of 60 Gray) plus Temozolomide 75 milligrams per square meter (mg/m2) capsules continuous daily oral dosing. In the maintenance phase after RT, patients stopped TMZ for 4 weeks and restarted TMZ at 150 mg/m2 in cycle 1 and 200 mg/m2 in cycles 2 to 6 on days 1 to 5 of 28-day treatment cycles. Patients were administered Afatinib 40 milligram (mg) film-coated tablet once daily after RT. Dose reductions of Afatinib were allowed if 40 mg or 30 mg were not tolerated. The treatment duration was until tumour progression or occurrence of undue adverse reactions, whichever occurred first.
- Afatinib 20 mg, Radiotherapy - Regimen U: Patients were administered Afatinib 20 mg film-coated tablet once daily orally plus radiotherapy (RT) i.e. focal radiation at a dose of 2 Gray per fraction on 5 days per week for 6 weeks (RT phase) (total dose of 60 Gray). Patients were administered Afatinib 40 milligram (mg) film-coated tablet once daily in the maintenance phase after RT. The treatment duration was until tumour progression or occurrence of undue adverse reactions, whichever occurred first. Dose reductions were allowed if 40 mg or 30 mg afatinib were not tolerated.
- Afatinib 40 mg, Radiotherapy - Regimen U: Patients were administered Afatinib 40 mg film-coated tablet once daily orally plus radiotherapy (RT) i.e. focal radiation at a dose of 2 Gray per fraction on 5 days per week for 6 weeks (RT phase) (total dose of 60 Gray). Patients were administered Afatinib 40 milligram (mg) film-coated tablet once daily in the maintenance phase after RT. The treatment duration was until tumour progression or occurrence of undue adverse reactions, whichever occurred first. Dose reductions were allowed if 40 mg or 30 mg afatinib were not tolerated.
Period: Overall Study
Arm/Group | Afatinib 20 Milligram, Radiotherapy + Temozolomide - Regimen M | Afatinib 30 mg, Radiotherapy + Temozolomide - Regimen M | Afatinib 40 mg, Radiotherapy + Temozolomide - Regimen M | Afatinib 20 mg, Radiotherapy - Regimen U | Afatinib 40 mg, Radiotherapy - Regimen U
Started | 7 | 6 | 7 | 3 | 13
Discontinued Afatinib Before/on Day 42 (Discontinued afatinib before or at the end of the concomitant treatment period (i.e. on day 42).) | 1 | 0 | 4 | 0 | 3
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 6 | 7 | 3 | 13
Not completed — Other than listed | 1 | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 4 | 0 | 6
Not completed — Dose-limiting toxicity (DLT) | 1 | 0 | 1 | 0 | 0
Not completed — Progressive disease | 2 | 6 | 1 | 3 | 5

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): Patients who received at least 1 dose of trial medication were included in the treated set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib 20 Milligram, Radiotherapy + Temozolomide - Regimen M | Afatinib 30 mg, Radiotherapy + Temozolomide - Regimen M | Afatinib 40 mg, Radiotherapy + Temozolomide - Regimen M | Afatinib 20 mg, Radiotherapy - Regimen U | Afatinib 40 mg, Radiotherapy - Regimen U | Total
Number analyzed (Participants) | 7 | 6 | 7 | 3 | 13 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Treated Set
  Years | 48.6 (15.7) | 52.7 (7.1) | 56.0 (9.1) | 52.0 (3.6) | 55.2 (9.3) | 53.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Treated Set
  Participants
    Female | 2 | 2 | 2 | 0 | 5 | 11
    Male | 5 | 4 | 5 | 3 | 8 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was not reported in this trial Population: Treated Set
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 1 | 0 | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0
    White | 7 | 5 | 7 | 3 | 13 | 35
    More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Investigator Defined Dose Limiting Toxicities (DLT) During the RT Phase
Description: Adverse event (AE) related to afatinib with any one criteria; Hematological: Common terminology criteria for adverse events (CTCAE) Grade 4 neutropenia (Absolute neutrophil count, including bands <500/cubic millimeter (mm³)) for >7 days, CTCAE Grade 3 or 4 neutropenia of any duration associated with fever >38.3 Celsius, CTCAE Grade 3 thrombocytopenia (platelet count <50000 - 25000/mm³), All other toxicities of CTCAE Grade ≥3 leading interruption of treatment > 14 days.
  Non-hematological: CTCAE Grade ≥3 nausea or vomiting despite appropriate use of standard anti-emetics for ≥3 days, CTCAE Grade ≥3 diarrhea despite appropriate use of standard anti-diarrheal therapy for ≥3 days, CTCAE Grade ≥3 rash despite standard medical management and lasting >7 days, CTCAE Grade ≥2 cardiac left ventricular function, CTCAE Grade ≥2 worsening of renal function as measured by serum creatinine, newly developed proteinuria or decrease in glomerular filtration rate, All other toxicities of CTCAE Grade ≥3.
Time Frame: 6 weeks
Population: Treated Set (TS); 3 patients were not evaluable for the determination of the maximum tolerated dose replaced in regimen M. 7 patients were excluded from the Afatinib 40 mg arm regimen U count as these were part of the expansion phase after the Maximum Tolerated Dose (MTD) had been determined.
Measure: Number; unit: Participants
Arm/Group | Afatinib 20 Milligram, Radiotherapy + Temozolomide - Regimen M | Afatinib 30 mg, Radiotherapy + Temozolomide - Regimen M | Afatinib 40 mg, Radiotherapy + Temozolomide - Regimen M | Afatinib 20 mg, Radiotherapy - Regimen U | Afatinib 40 mg, Radiotherapy - Regimen U
Number analyzed (Participants) | 6 | 6 | 5 | 3 | 6
Participants | 1 | 0 | 2 | 0 | 1

2. Secondary Outcome: Incidence and Intensity of Adverse Events (AE) According to Common Terminology Criteria of Adverse Events (CTCAE v.3.0)
Description: Incidence and intensity of adverse events (AE) according to Common Terminology Criteria of Adverse Events (CTCAE v.3.0). The CTCAE grades are: 1 (mild AE), 2 (moderate AE), 3 (severe AE), 4 (life-threatening or disabling AE), 5 (death related to AE).
Time Frame: From the first administration of trial medication until 4 weeks after the last administration of trial medication, up to approximately 338 weeks
Population: Treated Set
Measure: Number; unit: Participants
Arm/Group | Afatinib 20 Milligram, Radiotherapy + Temozolomide - Regimen M | Afatinib 30 mg, Radiotherapy + Temozolomide - Regimen M | Afatinib 40 mg, Radiotherapy + Temozolomide - Regimen M | Afatinib 20 mg, Radiotherapy - Regimen U | Afatinib 40 mg, Radiotherapy - Regimen U
Number analyzed (Participants) | 7 | 6 | 7 | 3 | 13
Participants
  Grade 1 | 0 | 0 | 1 | 0 | 1
  Grade 2 | 0 | 2 | 1 | 1 | 2
  Grade 3 | 4 | 4 | 4 | 2 | 5
  Grade 4 | 3 | 0 | 1 | 0 | 2
  Grade 5 | 0 | 0 | 0 | 0 | 3

3. Primary Outcome: Maximum Tolerated Dose (MTD) of Afatinib
Description: The MTD was defined as the highest afatinib dose level, at which no more than 1 out of 6 patients experienced drug-related DLT, i.e. the highest afatinib dose with a DLT incidence ≤17%. A separate MTD was determined for afatinib and RT (Regimen U), and for afatinib, TMZ, and RT (Regimen M).
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Number; unit: Milligram (mg)
Groups:
- Total - Regimen M: Patients were administered Afatinib 20/30/40 mg film-coated tablet once daily orally plus radiotherapy (RT) i.e. focal radiation at a dose of 2 Gray per fraction on 5 days per week for 6 weeks (RT phase) (total dose of 60 Gray) plus Temozolomide 75 milligrams per square meter (mg/m2) capsules continuous daily oral dosing. In the maintenance phase after RT, patients stopped TMZ for 4 weeks and restarted TMZ at 150 mg/m2 in cycle 1 and 200 mg/m2 in cycles 2 to 6 on days 1 to 5 of 28-day treatment cycles. Patients were administered Afatinib 40 milligram (mg) film-coated tablet once daily after RT. Dose reductions of Afatinib were allowed if 40 mg or 30 mg were not tolerated. The treatment duration was until tumour progression or occurrence of undue adverse reactions, whichever occurred first.
- Total - Regimen U: Patients were administered Afatinib 20/40 mg film-coated tablet once daily orally plus radiotherapy (RT) i.e. focal radiation at a dose of 2 Gray per fraction on 5 days per week for 6 weeks (RT phase) (total dose of 60 Gray). Patients were administered Afatinib 40 milligram (mg) film-coated tablet once daily in the maintenance phase after RT. The treatment duration was until tumour progression or occurrence of undue adverse reactions, whichever occurred first. Dose reductions were allowed if 40 mg or 30 mg afatinib were not tolerated.
Arm/Group | Total - Regimen M | Total - Regimen U
Number analyzed (Participants) | 17 | 9
Milligram (mg) | 30 | 40

4. Secondary Outcome: The Objective Tumour Response According to the Macdonald Criteria
Description: Objective response was defined as a best overall response of complete response (CR) or partial response (PR). The best overall response was the best overall response to trial medication according to the Macdonald criteria recorded since the first administration of trial medication and until the earliest of disease progression, death, or start of further anti-cancer treatment. Tumour response was assessed based on local radiological image evaluation by the investigators according to the Macdonald criteria: Complete Response (CR): Disappearance of all enhancing tumour on consecutive Magnetic resonance imaging (MRI) scans at least 28 days apart, off steroids, and neurologically stable or improved. Partial Response (PR): At least 50% reduction in size of enhancing tumour on consecutive MRI scans at least 28 days apart, steroids stable or reduced, and neurologically stable or improved.
Time Frame: as for outcome 2
Population: Treated Set
Measure: Number; unit: Participants
Arm/Group | Afatinib 20 Milligram, Radiotherapy + Temozolomide - Regimen M | Afatinib 30 mg, Radiotherapy + Temozolomide - Regimen M | Afatinib 40 mg, Radiotherapy + Temozolomide - Regimen M | Afatinib 20 mg, Radiotherapy - Regimen U | Afatinib 40 mg, Radiotherapy - Regimen U
Number analyzed (Participants) | 7 | 6 | 7 | 3 | 13
Participants
  No | 5 | 3 | 5 | 3 | 10
  Yes | 2 | 3 | 0 | 0 | 1
  Missing | 0 | 0 | 2 | 0 | 2

5. Secondary Outcome: Concentration of Afatinib in Plasma at Steady State Pre-dose on Days 8, 15 and 29
Description: Concentration of afatinib in plasma at steady state pre-dose (Cpre,ss) on days 8, 15 and 29.
Time Frame: Pharmacokinetic blood sample were taken at 5 minutes before drug on days 8, 15 and 29 and 1, 3 and 6 hours after drug administration on day 15
Population: Treated Set; only evaluable patients were included in the pharmacokinetic analysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Afatinib 20 Milligram, Radiotherapy + Temozolomide - Regimen M | Afatinib 30 mg, Radiotherapy + Temozolomide - Regimen M | Afatinib 40 mg, Radiotherapy + Temozolomide - Regimen M | Afatinib 20 mg, Radiotherapy - Regimen U | Afatinib 40 mg, Radiotherapy - Regimen U
Number analyzed (Participants) | 7 | 6 | 7 | 3 | 13
nanograms per milliliter (ng/mL)
  Cpre, ss, 8: number analyzed (Participants) | 3 | 5 | 5 | 3 | 12
  Cpre, ss, 8 | 4.4 (40.2) | 10.7 (70.3) | 15.7 (32.8) | 4.9 (32.9) | 16.7 (40.2)
  Cpre, ss, 15: number analyzed (Participants) | 4 | 6 | 4 | 3 | 10
  Cpre, ss, 15 | 5.6 (55.1) | 9.6 (54.3) | 16.8 (59.5) | 4.4 (177.0) | 18.9 (35.5)
  Cpre, ss, 29: number analyzed (Participants) | 4 | 6 | 3 | 3 | 9
  Cpre, ss, 29 | 5.3 (92.0) | 17.8 (15.6) | 17.4 (56.1) | 5.0 (53.3) | 16.1 (40.7)

ADVERSE EVENTS:
Time Frame: From the first administration of trial medication until 4 weeks after the last administration of trial medication, up to approximately 338 weeks
Arm/Group | Afatinib 20 Milligram, Radiotherapy + Temozolomide - Regimen M | Afatinib 30 mg, Radiotherapy + Temozolomide - Regimen M | Afatinib 40 mg, Radiotherapy + Temozolomide - Regimen M | Total - Regimen M | Afatinib 20 mg, Radiotherapy - Regimen U | Afatinib 40 mg, Radiotherapy - Regimen U | Total - Regimen U
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/7 | 0/20 | 0/3 | 3/13 | 3/16
Serious Adverse Events (participants affected / at risk) | 4/7 | 5/6 | 3/7 | 12/20 | 2/3 | 10/13 | 12/16
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 6/7 | 19/20 | 3/3 | 13/13 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 20 Milligram, Radiotherapy + Temozolomide - Regimen M (N=7) | Afatinib 30 mg, Radiotherapy + Temozolomide - Regimen M (N=6) | Afatinib 40 mg, Radiotherapy + Temozolomide - Regimen M (N=7) | Total - Regimen M (N=20) | Afatinib 20 mg, Radiotherapy - Regimen U (N=3) | Afatinib 40 mg, Radiotherapy - Regimen U (N=13) | Total - Regimen U (N=16)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Malaise (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 1
Meningitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 1 | 0 | 2 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 2
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 3
Seizure (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 2
Status epilepticus (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 20 Milligram, Radiotherapy + Temozolomide - Regimen M (N=7) | Afatinib 30 mg, Radiotherapy + Temozolomide - Regimen M (N=6) | Afatinib 40 mg, Radiotherapy + Temozolomide - Regimen M (N=7) | Total - Regimen M (N=20) | Afatinib 20 mg, Radiotherapy - Regimen U (N=3) | Afatinib 40 mg, Radiotherapy - Regimen U (N=13) | Total - Regimen U (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1 | 2 | 7 | 0 | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Ear pruritus (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diplopia (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1
Eye pain (Eye disorders) | 2 | 0 | 0 | 2 | 1 | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 2 | 1 | 6 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 5 | 5 | 17 | 3 | 11 | 14
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 6 | 4 | 5 | 15 | 1 | 2 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 1 | 2 | 3
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2 | 4 | 9 | 0 | 2 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 5 | 4 | 2 | 11 | 3 | 6 | 9
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Mucosal inflammation (General disorders) | 2 | 0 | 0 | 2 | 0 | 1 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Oedema peripheral (General disorders) | 1 | 0 | 1 | 2 | 0 | 1 | 1
Pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Unevaluable event (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 2 | 2
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1 | 1
Ear infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Localised infection (Infections and infestations) | 1 | 1 | 0 | 2 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 2 | 0 | 4 | 4
Nail bed infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 3 | 3
Paronychia (Infections and infestations) | 1 | 0 | 2 | 3 | 1 | 3 | 4
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Skin infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 2 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 3 | 0 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 3 | 0 | 3 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0 | 3 | 0 | 4 | 4
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 2 | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 1 | 3 | 0 | 1 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Escherichia test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Grip strength decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 2 | 0 | 0 | 2 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
QRS axis abnormal (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
White blood cells urine (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 1 | 4 | 0 | 1 | 1
Diet refusal (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 1 | 2 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 0 | 4 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 3 | 0 | 0 | 3 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Clumsiness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 0 | 1 | 3 | 0 | 1 | 1
Headache (Nervous system disorders) | 3 | 2 | 1 | 6 | 3 | 7 | 10
Hemianopia homonymous (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 4 | 5
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Neurological symptom (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 2
Partial seizures (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 3 | 0 | 0 | 3 | 1 | 2 | 3
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Speech disorder (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Mood altered (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1
Personality change (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Bladder pain (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1
Incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1
Orchitis noninfective (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Perineal erythema (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 0 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0 | 3 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 3 | 3 | 10 | 2 | 6 | 8
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 1 | 1 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 3 | 1 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 3 | 1 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 5 | 3 | 13 | 2 | 10 | 12
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 3 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/31/NCT00977431/Prot_000.pdf
  • Statistical Analysis Plan (2011-12-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT00977431/SAP_001.pdf